CLINICAL TRIAL: NCT02827071
Title: Ocular Imaging Study Using Advanced OCT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Steven Schwartz, Chief, Retina Division, University of California, Los Angeles
Other Study IDs: JSEI Nidek Advanced OCT
Record Dates: First submitted 2016-07-06; First posted 2016-07-11 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Retinal Vascular Disorder; Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Retina abnormalities: Subjects with various retina vascular disorders

SUMMARY:
The purpose of this study is to evaluate this AngioScan angiography software on patients with various retinal vascular disorders. The advanced OCT instrument is an FDA approved clinically used camera, but the AngioScan angiography software is not FDA approved. Investigators would like to know if this imaging device and software can improve the quality of images and visualization of imaged tissues and whether they are useful in the diagnosis and treatment of eye diseases. Images collected in this study may be compared to other images collected as part of standard of care on the same patient (OCT, FA, AF, Fundus).

ELIGIBILITY:
Inclusion Criteria:

• Any patient with abnormal retinal findings as determined by investigators.

Exclusion Criteria:

* Those suffering from head, neck or other injury which makes them unable to position themselves in head restraint for imaging.
* Participants who are unable to maintain retinal fixation on a specified target.
* Participants unable to achieve sufficient pupil dilation and alignment stability for imaging to take place.
* Patients with media opacity which preclude high quality imaging.

Ages: 18 Years to 115 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with retinal vascular abnormalities
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Retinal vascular abnormalities imaged by OCT Angiography and en face analysis of macular disorders | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Stein Eye Institute/Geffen School of Medicine, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No